CLINICAL TRIAL: NCT06492486
Title: Glioma Adaptive Radiotherapy With Development of an Artificial Intelligence Workflow
Acronym: GLADIATOR
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Tata Memorial Centre (Other)
Responsible Party: Principal Investigator, Dr Archya Dasgupta, Assistant Professor, Radiation Oncology, Tata Memorial Centre
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 4384
Record Dates: First submitted 2024-07-02; First posted 2024-07-09 (Actual); Last update posted 2025-09-16 (Actual); Status verified 2025-09

CONDITIONS: Diffuse Glioma; Glioblastoma; Adaptive Radiotherapy; Artificial Intelligence
MeSH Terms: conditions — Glioblastoma

STUDY DESIGN:
Intervention Model Description: The proposed Phase II prospective study will be split into two strata: IDH-negative GBM (stratum A) and IDH-mutant glioma (astrocytoma or oligodendroglioma) needing radiotherapy (stratum B).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Stratum A (IDH-negative GBM) (Experimental): Adaptive radiotherapy
  Interventions: Radiation: Adaptive radiotherapy
- Stratum B (IDH-mutant astrocytoma or oligodendroglioma) (Experimental): Adaptive radiotherapy
  Interventions: Radiation: Adaptive radiotherapy

INTERVENTIONS:
Radiation: Adaptive radiotherapy — Volumetric and biological adaptive radiotherapy will be delivered based on interval imaging with MRI and PET scan during treatment.

SUMMARY:
Gliomas are common primary brain tumors in adults. Gliomas can be classified into different types based on tumor grade, histopathological features, and molecular characteristics. The common types of diffuse gliomas include glioblastoma, astrocytoma, and oligodendroglioma. The standard treatment for diffuse gliomas includes surgery followed by radiation and chemotherapy. As per standard institutional practice, a uniform dose of radiation is delivered to the disease area and MRI is done before and after the treatment. In this study, MRI and PET scan will be done before starting the treatment and standard dose of radiation will be delivered. The interval imaging will be done twice during the course of treatment with MRI and PET, followed by dose modifications. The CT, MRI, and PET will be combined. Based on PET imaging, specific dose will be altered and delivered to specific areas. Dose modification will be done with the help of artificial intelligence. Participant's assessment will be done at regular intervals.

Modifications in radiation plans are done based on the changes in disease seen in scans is likely to improve the accuracy of RT treatments. Dose modifications based on imaging to resistant areas will help achieve better tumor control, reduce treatment-related toxicities, precise delivery of the RT and adjusting doses to the organs at risk (OAR) and changes in disease leading to better treatment compliance. Creating an artificial intelligence framework in radiation oncology promises to improve quality of workflow, treatment planning and RT delivery.

The aim of the study is to develop an artificial intelligence workflow for treatment of glioma with adaptive radiotherapy. This study will be conducted in Tata Memorial Centre on a population of 60 patients for a duration of 2 years. The total study duration is 4 years.

DETAILED DESCRIPTION:
Glioblastoma multiforme (GBM) represents grade 4 diffuse gliomas accounting for the most common primary malignant central nervous system (CNS) tumors in adults . GBM is treated with radiotherapy (RT) and concurrent chemotherapy following maximal safe resection, with a median survival of approximately 15-18 months . GBM harbors significant intratumoral heterogeneity with areas of multiclonal and hypoxic areas rendering higher chances of disease relapse following standard RT .

Similarly, distinct compartments can be well appreciated on magnetic resonance imaging (MRI): enhancing tumor core (TC) with central necrotic areas and the peritumoral region (PTR), which consists of microscopic tumor infiltration and vasogenic edema . Similar to regions of radioresistant areas within the TC, the microscopic disease in the PTR plays a vital role in disease relapse . Other grade 2 and 3 diffuse gliomas include isocitrate dehydrogenase (IDH) mutant astrocytoma and oligodendroglioma . In the recent World Health Organization (WHO) classification of CNS tumors, molecular information is combined with histopathological information for integrated classification. IDH-wildtype tumors are further molecularly characterized and considered as GBM since the prognosis is shown to be dismal. Oligodendrogliomas are confirmed based on the presence of deletion of 1p19q chromosomal arms. Grade 2/3 diffuse gliomas are typically seen as tumors with T2-weighted hyperintense tumors. The treatment is similar to GBM, with maximal safe resection followed by radiation and concurrent and adjuvant chemotherapy.

Radiotherapy for Diffuse Gliomas Radiotherapy (RT) forms an integral role in the multimodality management of diffuse gliomas . Radiation is indicated in low-grade gliomas with high-risk features or high-grade gliomas following maximal safe resection . The radiation (RT) in diffuse gliomas in GBM is delivered using conformal techniques to the residual disease and cavity, called the gross tumor volume (GTV). The surrounding area is included in the clinical target volume (CTV) to treat areas of microscopic disease. For GBM, an expansion of 1.5 -2 cm is done from the GTV, which is identified as an enhancing area on T1c sequences to include areas of PTR (T2w hyperintensity) and edited from anatomical barriers like meninges and dural reflections . For IDH-mutant gliomas, the residual tumor and cavity (identified as T2w hyperintensity region) are included as GTV and further expansion of 5-10 mm is done to be included as CTV . The standard practice involves delivering a uniform dose of radiation to the planning target volume (PTV), which encompasses an isotropic margin expansion surrounding the CTV to account for set-up uncertainties. In GBM and IDHmutant high-grade astrocytoma, the total dose of 59.4-60 Gy is delivered over 6-7 weeks with 1.8-2 Gy per fraction. A relatively lower dose of radiation, in the range of 54.0-59.4 Gy, is delivered over 6-7 weeks using 1.8-2 Gy per fraction for oligodendrogliomas. As per the current paradigm, radiation is planned on computed tomography (CT) for dose computation and MRI for visualization of target volumes and organs at risk (OAR), done once before treatment, based on which fractionated radiation is delivered over 6- 7 weeks. Recent evidence with MRI undertaken during the course of treatment has demonstrated the changes in dynamics of the residual disease, surgical cavity, and also the OARs in a proportion of patients, suggesting that treatment is delivered based on imaging at a single time-point can lead to inaccuracies .Therefore, adaptive radiotherapy (ART) to modify radiation plans based on the spatial changes of the target volume and OAR is likely to improve the accuracy of RT treatments. Also, serial imaging during treatment can be used to identify areas of tumor or PTR showing refractory disease or vasogenic edema, with provisions for biological modifications of RT doses . The use of conformal radiation techniques like intensity-modulated radiotherapy (IMRT), volumetric modulated arc therapy (VMAT) can enable delivery of differential radiation doses precisely to different areas of the target volume, known as dose painting .Positron Emission Tomography (PET) Functional imaging with positron emission tomography (PET) has attained wide popularity in oncology in disease staging, identifying hypoxic areas, and guiding radiation planning . For gliomas, amino acid PET like O-(2-[18F] fluoroethyl) -L-tyrosine (FET) or Fluorodopa (F-DOPA) has been proven effective with areas of a higher tumor to white matter ratio, suggestive areas of active disease (19) . The use of PET scans during treatment can help identify areas refractory to RT, reflected by higher uptake of the radioisotope. Higher doses to such regions provide a window for biological adaption and can potentially improve control rates. Similarly, quantitative analysis of imaging (more popularly known as radiomics) can help differentiate areas of microscopic tumor from vasogenic edema in the PTR, which otherwise appears similar to conventional imaging . Artificial Intelligence The role of artificial intelligence in oncology is increasingly recognized, ranging from optimization of healthcare resource utilization and decision-making to quantitative image analysis for prognostication and the potential ability to serve as a noninvasive biomarker . The practice of contemporary radiation oncology heavily relies on the interaction of humans and machines in almost every treatment planning process, including contouring of target volumes, OAR, treatment-planning processes, and during treatment delivery. Creating an artificial intelligence framework in radiation oncology promises to improve workflow efficiency and accuracy and enable treatment planning and delivery rapidly and efficiently. The use of adaptive radiotherapy will be further facilitated using machine learning algorithms with appropriate identification of patients to be benefitted from volumetric or biological adaptation, autosegmentation of target/OAR, automated treatment planning, and biological modification based on spatial and temporal changes of quantitative imaging parameters. Standard institutional practice The standard institutional practice includes a dose of 59.4 Gy in 33 fractions over 6.5 weeks for patients with glioblastoma and 55.8 Gy in 31 fractions over 6 weeks for patients with oligodendroglioma. Concurrent temozolomide is used for all patients undergoing radiation at the dose of 75 mg/m 2 of body surface area during the course of radiation with weekly monitoring on blood counts. All radiation treatments are planned based on single time CT and MRI scan without any scheduled interval scans during radiation, and no adaptation is done. Adjuvant chemotherapy with temozolomide is started after 4 weeks of radiation completion at dose of 150 mg/m 2 for five days and repeated on monthly basis and dose escalated to 200 mg/m 2 if tolerating well and normal blood counts. As standard practice 6 and 12 cycles of temozolomide are scheduled for GBM and IDH-mutant glioma (astrocytoma and oligodendroglioma) respectively. After treatment completion clinical follow-up is scheduled every 3-6 months in the first 2 years and thereafter every 6-12 months for all the patients. Surveillance imaging is scheduled every 6-12 months in the first 5 years and thereafter on annual basis or interval imaging undertaken as prompted clinically.

ELIGIBILITY:
Inclusion Criteria:

* Histological diagnosis of diffuse glioma. Patients with IDH-negative GBM (stratum A) and IDH-mutant glioma (astrocytoma or oligodendroglioma) need radiotherapy (stratum B).

Age: 18-70 years. Karnofsky Performance Scale (KPS) ≥60

Exclusion Criteria:

* Multifocal or multicentric disease Not eligible for radical intent radiation. IDH status is unknown or uninterpretable (IHC or gene sequencing). Use of prior radiotherapy to the head-neck region or brain or chemotherapy. Contraindication/unable to undergo MRI or PET scan during radiation.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-11-30 (Estimated); Primary Completion 2028-07-30 (Estimated); Study Completion 2028-07-30 (Estimated)

PRIMARY OUTCOMES:
Proportion of patients undergoing volumetric and biological adaptation. Cumulative rate of symptomatic radionecrosis (RN) at 2 years. | 2 years
  Proportion of patients where modification of radiation plan was done.
Cumulative rate of symptomatic radionecrosis at 2 years | 4 years
  Patients developing symptomatic radionecerosis will be analyzed using Kaplan-Meier survival method.

SECONDARY OUTCOMES:
Progression free survival | 4 years
  Progression free survival will be analyzed using Kaplan Meier method.
Overall survival | 4 years
  Overall survival will be analyzed using Kaplan Meier method.

CONTACTS AND LOCATIONS:
Overall Officials: Archya Dasgupta, Principal Investigator — Tata Memorial Centre

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ostrom QT, Patil N, Cioffi G, Waite K, Kruchko C, Barnholtz-Sloan JS. CBTRUS Statistical Report: Primary Brain and Other Central Nervous System Tumors Diagnosed in the United States in 2013-2017. Neuro Oncol. 2020 Oct 30;22(12 Suppl 2):iv1-iv96. doi: 10.1093/neuonc/noaa200. PMID 33123732
- [Background] Stupp R, Mason WP, van den Bent MJ, Weller M, Fisher B, Taphoorn MJ, Belanger K, Brandes AA, Marosi C, Bogdahn U, Curschmann J, Janzer RC, Ludwin SK, Gorlia T, Allgeier A, Lacombe D, Cairncross JG, Eisenhauer E, Mirimanoff RO; European Organisation for Research and Treatment of Cancer Brain Tumor and Radiotherapy Groups; National Cancer Institute of Canada Clinical Trials Group. Radiotherapy plus concomitant and adjuvant temozolomide for glioblastoma. N Engl J Med. 2005 Mar 10;352(10):987-96. doi: 10.1056/NEJMoa043330. PMID 15758009
- [Background] Tan AC, Ashley DM, Lopez GY, Malinzak M, Friedman HS, Khasraw M. Management of glioblastoma: State of the art and future directions. CA Cancer J Clin. 2020 Jul;70(4):299-312. doi: 10.3322/caac.21613. Epub 2020 Jun 1. PMID 32478924
- [Background] Dirkse A, Golebiewska A, Buder T, Nazarov PV, Muller A, Poovathingal S, Brons NHC, Leite S, Sauvageot N, Sarkisjan D, Seyfrid M, Fritah S, Stieber D, Michelucci A, Hertel F, Herold-Mende C, Azuaje F, Skupin A, Bjerkvig R, Deutsch A, Voss-Bohme A, Niclou SP. Stem cell-associated heterogeneity in Glioblastoma results from intrinsic tumor plasticity shaped by the microenvironment. Nat Commun. 2019 Apr 16;10(1):1787. doi: 10.1038/s41467-019-09853-z. PMID 30992437
- [Background] Shukla G, Alexander GS, Bakas S, Nikam R, Talekar K, Palmer JD, Shi W. Advanced magnetic resonance imaging in glioblastoma: a review. Chin Clin Oncol. 2017 Aug;6(4):40. doi: 10.21037/cco.2017.06.28. PMID 28841802
- [Background] Lemee JM, Clavreul A, Menei P. Intratumoral heterogeneity in glioblastoma: don't forget the peritumoral brain zone. Neuro Oncol. 2015 Oct;17(10):1322-32. doi: 10.1093/neuonc/nov119. Epub 2015 Jul 22. PMID 26203067
- [Background] Louis DN, Perry A, Wesseling P, Brat DJ, Cree IA, Figarella-Branger D, Hawkins C, Ng HK, Pfister SM, Reifenberger G, Soffietti R, von Deimling A, Ellison DW. The 2021 WHO Classification of Tumors of the Central Nervous System: a summary. Neuro Oncol. 2021 Aug 2;23(8):1231-1251. doi: 10.1093/neuonc/noab106. PMID 34185076
- [Background] Weller M, van den Bent M, Preusser M, Le Rhun E, Tonn JC, Minniti G, Bendszus M, Balana C, Chinot O, Dirven L, French P, Hegi ME, Jakola AS, Platten M, Roth P, Ruda R, Short S, Smits M, Taphoorn MJB, von Deimling A, Westphal M, Soffietti R, Reifenberger G, Wick W. EANO guidelines on the diagnosis and treatment of diffuse gliomas of adulthood. Nat Rev Clin Oncol. 2021 Mar;18(3):170-186. doi: 10.1038/s41571-020-00447-z. Epub 2020 Dec 8. PMID 33293629
- [Background] Mohile NA, Messersmith H, Gatson NT, Hottinger AF, Lassman A, Morton J, Ney D, Nghiemphu PL, Olar A, Olson J, Perry J, Portnow J, Schiff D, Shannon A, Shih HA, Strowd R, van den Bent M, Ziu M, Blakeley J. Therapy for Diffuse Astrocytic and Oligodendroglial Tumors in Adults: ASCO-SNO Guideline. J Clin Oncol. 2022 Feb 1;40(4):403-426. doi: 10.1200/JCO.21.02036. Epub 2021 Dec 13. PMID 34898238
- [Background] Halasz LM, Attia A, Bradfield L, Brat DJ, Kirkpatrick JP, Laack NN, Lalani N, Lebow ES, Liu AK, Niemeier HM, Palmer JD, Peters KB, Sheehan J, Thomas RP, Vora SA, Wahl DR, Weiss SE, Yeboa DN, Zhong J, Shih HA. Radiation Therapy for IDH-Mutant Grade 2 and Grade 3 Diffuse Glioma: An ASTRO Clinical Practice Guideline. Pract Radiat Oncol. 2022 Sep-Oct;12(5):370-386. doi: 10.1016/j.prro.2022.05.004. Epub 2022 May 31. PMID 35902341
- [Background] Tseng CL, Stewart J, Whitfield G, Verhoeff JJC, Bovi J, Soliman H, Chung C, Myrehaug S, Campbell M, Atenafu EG, Heyn C, Das S, Perry J, Ruschin M, Sahgal A. Glioma consensus contouring recommendations from a MR-Linac International Consortium Research Group and evaluation of a CT-MRI and MRI-only workflow. J Neurooncol. 2020 Sep;149(2):305-314. doi: 10.1007/s11060-020-03605-6. Epub 2020 Aug 29. PMID 32860571
- [Background] Niyazi M, Andratschke N, Bendszus M, Chalmers AJ, Erridge SC, Galldiks N, Lagerwaard FJ, Navarria P, Munck Af Rosenschold P, Ricardi U, van den Bent MJ, Weller M, Belka C, Minniti G. ESTRO-EANO guideline on target delineation and radiotherapy details for glioblastoma. Radiother Oncol. 2023 Jul;184:109663. doi: 10.1016/j.radonc.2023.109663. Epub 2023 Apr 13. PMID 37059335
- [Background] Hassanzadeh C, Rudra S, Ma S, Brenneman R, Huang Y, Henke L, Abraham C, Campian J, Tsien C, Huang J. Evaluation of interim MRI changes during limited-field radiation therapy for glioblastoma and implications for treatment planning. Radiother Oncol. 2021 May;158:237-243. doi: 10.1016/j.radonc.2021.01.040. Epub 2021 Feb 13. PMID 33587967
- [Background] Stewart J, Sahgal A, Lee Y, Soliman H, Tseng CL, Detsky J, Husain Z, Ho L, Das S, Maralani PJ, Lipsman N, Stanisz G, Perry J, Chen H, Atenafu EG, Campbell M, Lau AZ, Ruschin M, Myrehaug S. Quantitating Interfraction Target Dynamics During Concurrent Chemoradiation for Glioblastoma: A Prospective Serial Imaging Study. Int J Radiat Oncol Biol Phys. 2021 Mar 1;109(3):736-746. doi: 10.1016/j.ijrobp.2020.10.002. Epub 2020 Oct 14. PMID 33068687
- [Background] Senkesen O, Tezcanli E, Abacioglu MU, Ozen Z, Cone D, Kucucuk H, Goksel EO, Arifoglu A, Sengoz M. Limited field adaptive radiotherapy for glioblastoma: changes in target volume and organ at risk doses. Radiat Oncol J. 2022 Mar;40(1):9-19. doi: 10.3857/roj.2021.00542. Epub 2022 Mar 28. PMID 35368196
- [Background] Glide-Hurst CK, Lee P, Yock AD, Olsen JR, Cao M, Siddiqui F, Parker W, Doemer A, Rong Y, Kishan AU, Benedict SH, Li XA, Erickson BA, Sohn JW, Xiao Y, Wuthrick E. Adaptive Radiation Therapy (ART) Strategies and Technical Considerations: A State of the ART Review From NRG Oncology. Int J Radiat Oncol Biol Phys. 2021 Mar 15;109(4):1054-1075. doi: 10.1016/j.ijrobp.2020.10.021. Epub 2020 Oct 24. PMID 33470210
- [Background] Bentzen SM, Gregoire V. Molecular imaging-based dose painting: a novel paradigm for radiation therapy prescription. Semin Radiat Oncol. 2011 Apr;21(2):101-10. doi: 10.1016/j.semradonc.2010.10.001. PMID 21356478
- [Background] Galldiks N, Lohmann P, Albert NL, Tonn JC, Langen KJ. Current status of PET imaging in neuro-oncology. Neurooncol Adv. 2019 May 28;1(1):vdz010. doi: 10.1093/noajnl/vdz010. eCollection 2019 May-Dec. PMID 32642650
- [Background] Galldiks N, Niyazi M, Grosu AL, Kocher M, Langen KJ, Law I, Minniti G, Kim MM, Tsien C, Dhermain F, Soffietti R, Mehta MP, Weller M, Tonn JC. Contribution of PET imaging to radiotherapy planning and monitoring in glioma patients - a report of the PET/RANO group. Neuro Oncol. 2021 Jun 1;23(6):881-893. doi: 10.1093/neuonc/noab013. PMID 33538838
- [Background] Chaddad A, Kucharczyk MJ, Daniel P, Sabri S, Jean-Claude BJ, Niazi T, Abdulkarim B. Radiomics in Glioblastoma: Current Status and Challenges Facing Clinical Implementation. Front Oncol. 2019 May 21;9:374. doi: 10.3389/fonc.2019.00374. eCollection 2019. PMID 31165039
- [Background] Beig N, Bera K, Tiwari P. Introduction to radiomics and radiogenomics in neuro-oncology: implications and challenges. Neurooncol Adv. 2021 Jan 23;2(Suppl 4):iv3-iv14. doi: 10.1093/noajnl/vdaa148. eCollection 2020 Dec. PMID 33521636
- [Background] Dasgupta A, Geraghty B, Maralani PJ, Malik N, Sandhu M, Detsky J, Tseng CL, Soliman H, Myrehaug S, Husain Z, Perry J, Lau A, Sahgal A, Czarnota GJ. Quantitative mapping of individual voxels in the peritumoral region of IDH-wildtype glioblastoma to distinguish between tumor infiltration and edema. J Neurooncol. 2021 Jun;153(2):251-261. doi: 10.1007/s11060-021-03762-2. Epub 2021 Apr 27. PMID 33905055
- [Background] Huynh E, Hosny A, Guthier C, Bitterman DS, Petit SF, Haas-Kogan DA, Kann B, Aerts HJWL, Mak RH. Artificial intelligence in radiation oncology. Nat Rev Clin Oncol. 2020 Dec;17(12):771-781. doi: 10.1038/s41571-020-0417-8. Epub 2020 Aug 25. PMID 32843739